CLINICAL TRIAL: NCT07089329
Title: Efficacy of Striatin on Weight Gain, Improvement of Acute Phase Inflammatory Marker, and the Change of Firmicutes Bacteroidetes (F/B), SCFA, BDNF Proteins in Malnourished Children: A Preliminary Study
Brief Title: Efficacy of Striatin in Malnourished Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Collaborators: Dexa Medica Group (Industry)
Responsible Party: Principal Investigator, Moretta Damayanti Fauzi, MD, Child Health Department of Mohammad Hoesin Hospital, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University of Sriwijaya
Record Dates: First submitted 2025-06-17; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Severe Acute Malnutrition
Keywords: Striatin; Malnutrition; Acute inflammation markers; Microbiota; Children
MeSH Terms: conditions — Severe Acute Malnutrition; Malnutrition

STUDY DESIGN:
Intervention Model Description: It is a double-blind randomized controlled clinical trial to identify the effects of Striatin supplementation on weight, acute inflammation markers, and microbiota profiles of SAM children.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We use block randomization (http://www.randomization.com) to allocate the participants into intervention or placebo. The participants will receive a sequentially-numbered, opaque, sealed envelope (SNOSE) which each sealed envelope is given a sequential number according to the order of recruitment and it contains the randomization code. Pharmacists are responsible for the distribution of the SNOSE and intervention products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Striatin (Experimental): Participant in the intervention group will consume 1 sachet of the study product daily for 14 days. Each sachet contains 5 g of Striatin extract and 0.25 g of curcumin, to be dissolved in 10 ml of solvent syrup. The product is white in powder form, has sweet taste, and turns into a light-orange liquid after dissolution.
  Interventions: Drug: Striatin
- Placebo (Placebo Comparator): Participant in the control group will consume 1 sachet of Placebo daily for 14 days. Each sachet contains 4.89 g Mannitol, also to be dissolved in 10 ml of solvent syrup. The color and taste of the placebo match those of the intervention product to maintain blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Striatin — Daily administration of Striatin extract will be carried out for 14 days. The dose is 1 sachet/day (5 g of Striatin) which dissolved in 10 mll of syrup.
  Other Names: Inbumin Forte
  Arms: Striatin
Drug: Placebo — Daily administration of 1 sachet of placebo will be carried out for 14 days.
  Arms: Placebo

SUMMARY:
This is a double-blind randomized-controlled clinical trial to identify the effect of Striatin (snakehead fish extract) supplementation in increasing body weight, improving acute inflammatory markers and microbiota profiles in children with severe acute malnutrition (SAM) treating with standard nutritional therapy.

The main questions to answer are:

Does Striatin supplementation effective in increasing body weight and improving acute inflammatory markers in SAM children? What are the adverse events of Striatin supplementation in SAM children?

Researchers will compare Striatin supplementation and placebo (a look-alike substance that contains no drug) to identify the increase of body weight, improvement of acute inflammatory markers and microbiota profiles.

DETAILED DESCRIPTION:
1. Children aged 12-59 months diagnosed with SAM based on weight-for-height Z score (WHZ) and/or mid-upper arm circumference (MUAC) will be included in the study.
2. Informed consents will be given and drawn from mother or legal caregiver.
3. Blood and stool samples will be taken before and after intervention in all participants. Markers which will be checked are: prealbumin, hsCRP, and brain-derived neurotropic factor (BDNF), from blood. Moreover, short-chain fatty acid (SCFA) and Bacteroides/Firmiculates ratio will be analyzed from stool.
4. Block randomization will be conducted to allocate participants into two groups: intervention group who receive Striatin supplementation, and control group who receive placebo.
5. The intervention will be given for 14 days. Neither researchers nor participants aware of the type of intervention (Striatin or placebo).
6. Both groups will receive standard F-100 formula or oral nutrition therapy (ONS) as nutritional treatment for SAM, vitamin C, vitamin B complex, and folic acid.
7. Intervention group will receive 1 sachet of Striatin and control group will receive 1 sachet of Placebo every 24 hours. Both Striatin and placebo will be dissolved in 10 ml of solvent syrup. The route of administration can be oral or via nasogastric tube.
8. Weight will be measured every three days, and any complaint or side effect that appeared will be recorded every day.

ELIGIBILITY:
Inclusion Criteria:

1. Severe acute malnutrition (SAM) children based on WHZ and/or MUAC
2. Consents are given by parents/caregivers.

Exclusion Criteria:

1. SAM children with malignancy, liver cirrhosis, acute liver failure, severe kidney disorders, acute and chronic infections that attack the liver or other severe infections that require special treatment.
2. Subjects who require special anthropometric examinations (condition such as edema, organomegaly, amputation, cerebral palsy GMFCS > 2)
3. Children who have history of severe hypersensitivity to snakehead fish and/or cow's milk.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Absolute and relative weight increase | Baseline, every three days, and Day 15.
  Weight in grams
The change of Prealbumin | Baseline and Day 15.
  Prealbumin level
The change of hsCRP | Baseline and Day 15.
  hsCRP level

SECONDARY OUTCOMES:
The change of SCFA | Baseline and Day 15.
  Short chain fatty acids (SCFA)
The change ofB/F ratio | Baseline and Day 15.
  Bacteroides-Firmicutes ratio (B/F ratio)
Level of neurocognitive biomarker. | Baseline and Day 15.
  Brain Derived Neurotropic Factor (BDNF)

CONTACTS AND LOCATIONS:
Overall Officials: Agrifina Helga, Bachelor, Study Director — University of Sriwijaya
Locations (1):
- Community Health Center and Pediatric outpatient clinic at Mohammad Hoesin Hospital, Palembang, South Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sigh S, Roos N, Chamnan C, Laillou A, Prak S, Wieringa FT. Effectiveness of a Locally Produced, Fish-Based Food Product on Weight Gain among Cambodian Children in the Treatment of Acute Malnutrition: A Randomized Controlled Trial. Nutrients. 2018 Jul 16;10(7):909. doi: 10.3390/nu10070909. PMID 30012981
- [Background] Puji Rahayu, Faustine Marcelline, Erna Sulistyaningrum, Maggy Thenawidjaja Suhartono, Raymond Rubianto Tjandrawinata, Potential effect of striatin (DLBS0333), a bioactive protein fraction isolated from Channa striata for wound treatment, Asian Pacific Journal of Tropical Biomedicine, Volume 6, Issue 12, 2016, Pages 1001-1007, ISSN 2221-1691, https://doi.org/10.1016/j.apjtb.2016.10.008. (https://www.sciencedirect.com/science/article/pii/S2221169115308534)